CLINICAL TRIAL: NCT00053326
Title: A Phase II Study of Fenretinide (NSC# 374551, IND# 40294) in Children With Recurrent/Resistant High Risk Neuroblastoma
Brief Title: Fenretinide in Treating Children With Recurrent or Resistant Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01802; NCI-2012-01802 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL0024; COG-A0996; CDR0000269408; COG-ANBL0321; ADVL0024 (Other: Children's Oncology Group); ANBL0321 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: Recurrent Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Fenretinide

ARMS (1):
- Treatment (fenretinide) (Experimental): Patients receive oral fenretinide 3 times daily (or 2 times daily if over 18 years of age) on days 1-7. Treatment repeats every 3 weeks for up to 30 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fenretinide; Other: pharmacological study

INTERVENTIONS:
Drug: fenretinide — Given orally
Other: pharmacological study — Optional correlative studies

SUMMARY:
This phase II trial is studying how well fenretinide works in treating children with recurrent or resistant neuroblastoma. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

Determine the response rate in pediatric patients with recurrent or resistant high-risk neuroblastoma treated with fenretinide.

Determine the toxic effects of this drug in these patients. Determine the proportion of patients with disease detected only by bone marrow immunocytology, who clear all evidence of disease during treatment with this drug.

Determine minimal residual disease response by marrow and meta-iodobenzylguanidine (MIBG) I 123 scan in patients treated with this drug.

OUTLINE: Patients are stratified according to presence of measurable disease on CT scan/MRI (yes vs no). A third stratum of patients with tumor cells in bone marrow by immunocytology only is enrolled but is not evaluated for response.

Patients receive oral fenretinide 3 times daily (or 2 times daily if over 18 years of age) on days 1-7. Treatment repeats every 3 weeks for up to 30 courses in the absence of disease progression or unacceptable toxicity. Patients in stratum III who fail to achieve a complete response after 8 courses of therapy are removed from study.

Patients are followed monthly until blood counts and visual acuity are stable or normalized and then every 6 months for 2 years and annually for 3 years.

PROJECTED ACCRUAL: A total of 70 patients (25 each for strata I and II, 20 for stratum III) will be accrued for this study within 1-2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent or resistant/refractory high-risk neuroblastoma by one or both of the following:

  * Histological confirmation
  * Demonstration of tumor cells in bone marrow with increased urinary catecholamines
* Stratum I:

  * At least 1 unidimensionally measurable lesion*

    * At least 20 mm by MRI and/or CT scan OR at least 10 mm by spiral CT scan
* Stratum II: Meets one or both of the following criteria:

  * At least 1 site with positive uptake on meta-iodobenzylguanidine (MIBG) I 123 scan
  * Tumor in bilateral bone marrow aspirate/biopsy by routine morphology (no NSE staining only)
* Stratum III:

  * At least 5 tumor cells/10^6 mononuclear cells in the bone marrow by immunocytology only (on 2 successive bone marrows performed from 1 day to 4 weeks apart)
* Patients in first response (i.e., patients with persistent tumor at end of frontline therapy, but who have never had disease relapse or progression) must have histological* or morphological (by bone marrow) confirmation** of viable tumor on CT scan, MRI, or MIBG scan after completion of myeloablative therapy (for strata I and II)
* No catecholamine elevation only
* Performance status - 0-2
* At least 2 months
* Hemoglobin greater than 7.5 g/dL (transfusion allowed)
* Bilirubin no greater than 1.5 times normal
* SGPT and SGOT less than 2.5 times normal
* Creatinine normal for age
* No hematuria or proteinuria greater than 1+ on urinalysis
* Calcium less than 11.6 mg/dL
* Triglycerides less than 300 mg/dL
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No seizure disorders unless on anticonvulsants and well controlled
* No skin toxicity greater than grade 1
* Must be able to consume entire intact study capsule in the dosage prescribed for body surface area
* Recovered from prior immunotherapy
* At least 7 days since prior anticancer biologic therapy
* At least 2 days since prior growth factors
* Prior autologous stem cell transplantation allowed
* No prior allogeneic stem cell transplantation
* No concurrent immunomodulating agents
* At least 2 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* No concurrent anticancer chemotherapy
* No concurrent steroids
* Recovered from prior radiotherapy
* At least 4 weeks since prior radiotherapy to target lesion
* Prior radiotherapy to non target lesions allowed
* No concurrent radiotherapy to sole measurable lesion for symptom relief
* Concurrent palliative radiotherapy to non target or localized painful lesions allowed
* Prior tretinoin or isotretinoin allowed
* At least 2 weeks since other prior retinoids
* No prior fenretinide
* No concurrent supplemental oral or IV vitamin A, ascorbic acid, or vitamin E (except if contained in routine total parenteral nutrition [TPN] vitamin supplements)
* No concurrent drugs suspected of causing pseudotumor cerebri (e.g., tetracycline, nalidixic acid, nitrofurantoin, phenytoin, sulfonamides, lithium, amiodarone, or vitamin A [except as part of routine TPN supplements])
* No other concurrent anticancer agents

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2003-05; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 8 courses of therapy
  A responder is defined to be a patient who achieves a best overall response of complete response (CR), very good partial response (VGPR) or partial response (PR).
Toxicity as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 5 years
  Assessed via a descriptive tabulation of the toxicity rates, overall and by stratum.

SECONDARY OUTCOMES:
Levels of fenretinide | At baseline and during courses 1, 2, and 5
  Assessed via descriptive analysis of the steady state levels of fenretinide overall and by stratum
Plasma retinol levels | At baseline and during courses 1, 2, and 5
  Assessed via descriptive analysis of the plasma retinol levels overall and by stratum.
Minimal residual disease (MRD) (Stratum 3) | Up to 5 years
  Assessed by descriptive calculation of the proportion of responders.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Villablanca, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States